The Effect of Self-Compassion Based Birth Preparation Program on Self-Compassion, Body Image, Fear of Childbirth, Depression, Anxiety and Stress in Pregnant Women

## INFORMED CONSENT FORM

## Dear Participant,

I am Hilal Gül BOYRAZ YANIK, a PhD student at Ordu University Health Sciences Institute, Department of Obstetrics and Gynecology Nursing. I am conducting a PhD thesis titled "The Effect of Self-Compassion Based Birth Preparation Program on Self-Compassion, Body Image, Fear of Childbirth, Depression, Anxiety and Stress in Pregnant Women". The findings obtained in line with the answers you will sincerely give during the study will contribute to determining the effect of self-compassion based birth preparation program during pregnancy on self-compassion, body image, fear of childbirth, depression, anxiety and stress.

Self-compassion training in the study will be given to you by the researcher Res. Asst. Hilal Gül BOYRAZ YANIK. The program is planned to last 8 sessions. Necessary permissions have been obtained for the study. The study does not include any intervention other than the hospital procedure you are currently in and does not carry any risks.

A questionnaire and scales will be applied to you regarding our study topic. If there is any development that may concern you during the study, you will be notified. Participation in this study is entirely voluntary. You may refuse to participate in the study or withdraw from the study at any stage. This will not prevent your benefits. The results of the study will be used for scientific purposes; if you withdraw from the study or are removed by the researcher, your medical data may also be used for scientific purposes if necessary.

All your medical and identity information will be kept confidential and your identity information will not be disclosed even if the study is published, but the audience of the study, those conducting the examination, ethics committees and official authorities may access your medical information when necessary. You may also access your own medical information if you wish.

## **Consent to Participate in the Study:**

I have read and verbally listened to the information provided above, which should be given to the volunteer before the study begins. I have asked the researcher all the questions that come to my mind, and I have fully understood all the written and verbal explanations given to me. I have been given sufficient time to decide whether I want to participate in the study. Under these conditions, I authorize the researcher to review, transfer and process my medical information and I accept the invitation to participate in this research voluntarily, without any coercion or pressure. A signed copy of this form will be given to me.

Volunteer's,

Name-Surname:

Address:

Tel.-Fax:

Date and Signature: The researcher who made the statements,

Name-Surname: Hilal Gül BOYRAZ

YANIK

Position: Research Assistant

Address: Ordu University Faculty of Health

Sciences Tel.-Fax:

Date and Signature: